CLINICAL TRIAL: NCT05053919
Title: Sleep Improvement of Schumann Resonance in the Treatment of Insomnia-A Randomized and Double-blinded Study
Brief Title: Schumann Resonance and Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101267B0
Record Dates: First submitted 2021-08-06; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Insomnia
Keywords: Insomnia; Schumann resonance; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SR device group (Experimental)
  Interventions: Device: Schumann resonance sleep device
- placebo device group (Placebo Comparator)
  Interventions: Device: Placebo sleep device

INTERVENTIONS:
Device: Schumann resonance sleep device — A Schumann resonance sleep device would stably output the composite frequency of a "the Schumann resonance frequency (7.83 Hz) wave, theta wave, and delta wave".
  The subjects were asked to use the device (place it next to the bed facing the subject's head, turn it on about one hour before going to bed every night, and turn it off after getting up the next day) every night for four weeks.
  Arms: SR device group
Device: Placebo sleep device — A Placebo sleep device is an instrument with the same appearance and operation as the Schumann resonance sleep device, but does not output any frequency wave.
  The subjects were asked to use the device (place it next to the bed facing the subject's head, turn it on about one hour before going to bed every night, and turn it off after getting up the next day) every night for four weeks.
  Arms: placebo device group

SUMMARY:
The double-blinded and randomized study evaluated the effectiveness and side effects of a novel non-invasive treatment, Schumann resonance (SR), in treating insomnia. The objective of this study is (1) to evaluate the improvement of sleep quality of patients with insomnia disorder by SR and (2) to be the basis for the future development of physical magnetic therapy.

DETAILED DESCRIPTION:
Insomnia is a common sleep disturbance that affects the health and quality of life of individuals and accounts for considerable utilization of medical resources. The prevalence of insomnia is approximately 30%; in Asia, the prevalence of insomnia is approximately 4% in Japan, 9.9% in South Korea, 10.3% in Taiwan. Based on the statistic of Taiwan BNHI office in a 2013 report, there is worth of 1.3 billion prescriptions of hypnotic drug in one year. In addition, the reimbursement expenditure pays up more than 1 billion New Taiwan Dollars (NTD) with increasing expense rate of 15% every year, showing insomnia causes great distress to Taiwanese.

The characteristics of insomnia are difficulty with initiating or maintaining sleep, early morning waking, or non-restorative sleep. In DSM-5, the diagnosis of primary insomnia has been renamed insomnia disorder to avoid the differentiation between primary and secondary insomnia.

The most common treatment for insomnia is pharmacological therapy with hypnotics such as a benzodiazepine, zolpidem, or zopiclone. However, treatment with hypnotics includes the risk of adverse effects, drug tolerance and dependence . Some past reports on different non-pharmacological treatment strategies, such as Cognitive-Behavioral Therapy (CBT), muscle relaxation training, stimulus control, sleep restriction, and sleep hygiene, have demonstrated the effectiveness of most of these non-pharmacological treatments. However, the poor compliance and inconvenience for CBT is always a big issue.

Except the traditional treatment of insomnia, some folk therapies' clinical effect does not been confirmed, such as aromatherapy, music therapy, etc. Nowadays, due to development of technology for medical devices, some sleep devices were launched, aim to prolong the slow-wave sleep and enhances the sleeping quality.

The investigational device in this study is a sleep device with SRF (Sleep Restore Frequency), the principle is to integrate the bio-energy generated Schumann resonances, native from Earth, and the shocks from the Earth's magnetic field. Through the non-contact method with bio-energy waves, SRF are coupled to the sleep center of the brain, inducing and adjusting the electrical activities of the sleep center. It prolongs the in-depth sleep and enhances the sleeping quality.

The objective of this study is (1) to evaluate the improvement of sleep quality of patients with insomnia disorder by sleep device and (2) to be the basis for the future development of physical magnetic therapy.

Sample Size Approximately 60 subjects who meet the inclusion and exclusion criteria will be enrolled into the trial and averagely separated two arms for statistical analysis.

Statistical Analysis Efficacy evaluation statistics will be conducted with independent t-test or Fisher's exact test for testing the differences and conducted with Pearson correlation coefficient for the association between variables.

ELIGIBILITY:
Inclusion Criteria:

* (1) participants are between 20 and 70 years old;
* (2) participants must meet the DSM-5 diagnostic criteria for insomnia and have been diagnosed for more than three months;
* (3) participants must be willing to sign an informed consent form;
* (4) participants who took sleep aiding pills must cooperate not to change any medication and dosage during the study.

Exclusion Criteria:

* (1) participants using pacemakers or cardiac monitors;
* (2) participants with severe physical illness or after surgery, such as heart disease, metabolic diseases, or cancer;
* (3) participants with severe mental disorders, such as schizophrenia, severe major depression, severe anxiety, bipolar disorder, dementia, substance use disorder; or severe neurological diseases such as a seizure, stroke or Parkinson's disease;
* (4) participants with other serious sleep disorders, such as severe sleep obstructive apnea, severe periodic limb movement syndrome or narcolepsy;
* (5) participants who are unable to attend regular follow-up evaluations;
* (6) participants who are unable to keep good sleep hygiene and cannot stop using electronic products before going to bed.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-01-19 (Estimated); Study Completion 2022-01-19 (Estimated)

PRIMARY OUTCOMES:
actigraphy | 4 weeks
  Change in sleep latency (mins) based on actigraphy from before treatment to after treatment.

SECONDARY OUTCOMES:
actigraphy-TST | 4 weeks
  Total sleep time (TST, mins) based on actigraphy from before treatment to after treatment.
actigraphy-SE | 4 weeks
  Sleep efficiency (SE, %) based on actigraphy from before treatment to after treatment.
actigraphy-WASO | 4 weeks
  Wake after sleep onset (WASO) based on actigraphy from before treatment to after treatment.
polysomnography (PSG)-SL | before and after 4 weeks using sleep device
  Change in sleep latency (SL, mins) based on PSG from before treatment to after treatment.
polysomnography (PSG)-TST | before and after 4 weeks using sleep device
  Change in total sleep time (TST, mins) based on PSG from before treatment to after treatment.
polysomnography (PSG)-SE | before and after 4 weeks using sleep device
  Change in sleep efficiency (SE, %) based on PSG from before treatment to after treatment.
polysomnography (PSG)-WASO | before and after 4 weeks using sleep device
  Change in wake after sleep onset (WASO, mins) based on PSG from before treatment to after treatment.
polysomnography (PSG)-SWS | before and after 4 weeks using sleep device
  Change in slow wave sleep (SWS, %) based on PSG from before treatment to after treatment.
polysomnography (PSG)-REM | before and after 4 weeks using sleep device
  Change in REM sleep (%) based on PSG from before treatment to after treatment.
Pittsburgh Sleep Quality Index (PSQI) | before, after 2 weeks, and after 4 weeks using sleep device
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire for assessing the subjective sleep quality, which consists of 19 items and can be calculated and combined into 7 clinically-derived component score (0-3), with higher scores indicating worse sleep quality.
36-Item Short-Form Health Survey (SF-36) | before, after 2 weeks, and after 4 weeks using sleep device
  36-Item Short-Form Health Survey (SF-36) includes 11 major questions that evaluate eight components (0-100), with higher scores indicating better outcome.These components include physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional wellbeing, social functioning, pain, and general health.
sleep diary (sleep logs)-SL | before, after 2 weeks, and after 4 weeks using sleep device
  From the diaries, an estimate was computed for an average of sleep latency (SL, mins).
sleep diary (sleep logs)-TST | before, after 2 weeks, and after 4 weeks using sleep device
  From the diaries, an estimate was computed for an average of total sleep time (TST, mins).
sleep diary questionaire (sleep logs)-SE | before, after 2 weeks, and after 4 weeks using sleep device
  From the diaries, an estimate was computed for an average of sleep efficiency (SE, %).

OTHER OUTCOMES:
heart rate variability (HRV) device | before, after 2 weeks, and after 4 weeks using sleep device
  The measurement method is to stick four patches on participants body and measure the heart rhythm state for 10 minutes. An estimate was computed for LF/HF ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided